CLINICAL TRIAL: NCT00381576
Title: Multiple Sclerosis and Muscle Function - Effects of Heavy Progressive Resistance Training
Brief Title: Multiple Sclerosis and Heavy Progressive Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Sonderborg Hospital (Other Government); The Danish Multiple Sclerosis Society (Unknown)
Responsible Party: Department of sports science, Aarhus University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 300976
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Multiple Sclerosis
Keywords: Resistance training; Strength training; Training adaptations; CNS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): 12 weeks of resistance training
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — Intervention group: 12 weeks of resistance training for the lower extremity. Control group: No intervention - 12 weeks of normal daily living

SUMMARY:
The purpose of the present investigation is to determine whether MS patients can tolerate and benefit from heavy progressive resistance training. A second purpose is to determine both neural and muscle morphological adaptations to heavy progressive resistance training.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) patients are characterized by reduced muscle strength and functional capacity. For MS patients, improvements in muscle strength and thereby functional capacity, would have the potential to make both the daily living easier and to extend the time living independently. Attempts to improve muscle strength and function include the application of physical training, although the general advice to MS patients for many years has been to avoid participation in physical training. It has now been demonstrated that endurance training at low to moderate intensity is well tolerated by MS patients, but it only induces modest improvements in both muscle strength and functional capacity. Heavy progressive resistance training (HPRT) has proven to be the most effective means to improve muscle strength and functional capacity during daily activities in healthy older people. However, the effects of HPRT have not been investigated in randomised control trials in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Relapsing Remitting Multiple Sclerosis according to the McDonald criteria
* Expanded Disability Status Scale Score between 3,0-5,5
* Be able to walk at least 100m
* Be able to train twice a week at the University

Exclusion Criteria:

* Alcohol abuse, Alzheimer's and pacemaker
* Comorbidities like cardiovascular-, respiratory-, orthopaedic or metabolic diseases
* Having had an attack in a period of 8 weeks prior to the start of the intervention period
* Having an attack during the intervention period
* Pregnancy
* Systematic resistance training in a period of 3 months prior to the start of the intervention period.
* Training adherence of less than 85%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Muscle strength (isokinetic testing) | Before and after the intervention

SECONDARY OUTCOMES:
Functional capacity (Six minute walk test, 10m walk test, chair rise, stair climbing) | Before and after the intervention
Muscle biopsies from m. vastus lateralis | Before and after the intervention
% Fat (skinfold) | Before and after the intervention
Blood samples (immunologic parameters) | Before and after the intervention
Fatigue (Fatigue Severity Scale - FSS, Modified Fatigue Inventory - MFI-20) | Before and after the intervention
HRQOL: SF36 | Before and after the intervention
Depression: Major Depression Inventory (MDI) | Before and after the intervention
Surface EMG from m. vastus lateralis during MVC | Before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Dalgas, Ph.d. Stud., Principal Investigator — Department of Sports Science, University of Aarhus; Thorsten Ingemann-Hansen, Professor, Study Chair — Department of Sports Science, University of Aarhus; Egon Stenager, MD, Study Chair — MS clinic, Department of Neurology, Sonderborg Hospital
Locations (2):
- Denmark (2):
  - MS Clinic, Department of Neurology, Aarhus University Hospital, Aarhus
  - Department of Sports Science, University of Aarhus, Aarhus

REFERENCES:
- [Derived] Dalgas U, Stenager E, Lund C, Rasmussen C, Petersen T, Sorensen H, Ingemann-Hansen T, Overgaard K. Neural drive increases following resistance training in patients with multiple sclerosis. J Neurol. 2013 Jul;260(7):1822-32. doi: 10.1007/s00415-013-6884-4. Epub 2013 Mar 13. PMID 23483214
- [Derived] Dalgas U, Severinsen K, Overgaard K. Relations between 6 minute walking distance and 10 meter walking speed in patients with multiple sclerosis and stroke. Arch Phys Med Rehabil. 2012 Jul;93(7):1167-72. doi: 10.1016/j.apmr.2012.02.026. Epub 2012 Mar 12. PMID 22421626